CLINICAL TRIAL: NCT06982235
Title: Stone and Laser Therapies Post-Market Study
Brief Title: Stone and Laser Therapies Post-Market Study (SALT)
Acronym: SALT
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0777
Record Dates: First submitted 2025-04-30; First posted 2025-05-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Benign Prostate Hypertrophy(BPH); Renal Calculi; Ureteral Stones, Kidney Stones; Calculi, Urinary; Urinary Tract Procedure
Keywords: BPH; Benign Prostatic Hyperplasia; Lithotripsy; Renal Calculi; Renal Calculus; Boston Scientific; Kidney Stone; Urinary Tract Procedure
MeSH Terms: conditions — Prostatic Hyperplasia; Kidney Calculi; Urinary Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Urinary Tract Procedure Cohort: Subjects intend to undergo diagnostic and/or therapeutic urinary tract procedure with study device(s)
  Interventions: Device: Ureteroscope system; Device: Laser system
- Benign Prostatic Hyperplasia Cohort: Subjects are at least 40 years of age diagnosed with BPH with lower urinary tract symptoms and intend to undergo BPH treatment with study device(s)
  Interventions: Device: Laser system

INTERVENTIONS:
Device: Ureteroscope system — LithoVue™ Elite Single-Use Digital Flexible Ureteroscope System with intrarenal pressure monitoring
  Groups: Urinary Tract Procedure Cohort
Device: Laser system — Pulse™ 120H Holmium Laser System with MOSES™ 2.0 Technology

SUMMARY:
The objective of the SALT Study is to obtain post-market safety and device performance data for Boston Scientific's Stone and BPH study devices used during a diagnostic and/or therapeutic urinary tract procedure (e.g., transurethral or percutaneous access routes) or benign prostatic hyperplasia (BPH) treatment.

DETAILED DESCRIPTION:
The SALT study is a multi-center, open label, non-randomized, prospective observational study to document on-going post-market safety and device performance data of BSC commercially available study devices that are used in diagnostic and/or therapeutic urinary tract procedures or surgical treatment for BPH.

Enrolled subjects undergoing diagnostic or therapeutic procedures using study devices will be followed for 1 year after the index procedure is complete.

ELIGIBILITY:
Inclusion Criteria:

For urinary tract procedure cohort:

1. Subject intends to undergo diagnostic and/or therapeutic urinary tract procedure with qualified BSC device(s)
2. Subject is willing and able to complete all follow-up visits

For BPH cohort:

1. Subject is ≥ 40 years of age
2. Subject with a diagnosis of benign prostatic hyperplasia (BPH) with lower urinary tract symptoms
3. Subject intends to undergo BPH treatment with qualified BSC device(s)
4. Subject is willing and able to complete all follow-up visits

Exclusion Criteria:

For urinary tract procedure cohort:

1. Subject requires simultaneous surgical treatment for BPH
2. Unwilling or unable to provide consent
3. Any other condition which, in the opinion of the investigator, precludes study participation (e.g., history of medical non-compliance, etc.)

For BPH cohort:

1. Subject requires simultaneous upper urinary calculi lithotripsy procedure (not applicable to bladder calculi)
2. Unwilling or unable to provide consent
3. Any other condition which, in the opinion of the investigator, precludes study participation (e.g., history of medical non-compliance, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The SALT study will enroll subjects undergoing a diagnostic or therapeutic urinary tract procedure, or benign prostatic hyperplasia (BPH) procedure, using study devices. Subjects will generally be recruited from Investigators' practices. A minimum of 119 subjects will be enrolled in each cohort.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Serious Adverse Events related to BSC study devices | From procedure to 12-months after the procedure
  The primary endpoint is the occurrence of serious adverse events related to BSC study devices.

SECONDARY OUTCOMES:
Assess Stone Free Rate in therapeutic Urinary Tract Procedures | 21 - 90 days after the procedure
  For upper urinary tract stone procedures: Stone clearance assessed by stone free rate (SFR) at the post procedure imaging study.
Change in BPH symptoms | 6 months after the procedure
  In subjects with applicable benign prostatic hyperplasia (BPH) procedure(s): Improvement in BPH symptoms from baseline as measured by favorable change (decrease) in International Prostate Symptom Score (IPSS) at 6 months follow up, on a scale of 0 to 35.

OTHER OUTCOMES:
Health status as measured by EQ-5D-5L | From baseline through post-procedure standard-of-care follow-up within 12 months of the index procedure
  Pre-and post-operative health status as measured by a validated quality-of-life questionnaire, the EQ-5D five-level (5L) (EQ-5D-5L).
  The first part (the descriptive system) assesses health in five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT, ANXIETY / DEPRESSION), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to). This part of the EQ-5D questionnaire provides a descriptive profile that can be used to generate a health state profile. Each health state can potentially be assigned a summary index score based on societal preference weights for the health state. Health state index scores generally range from less than 0 to 1 (the value of full health), with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale (VAS) to rate perceived health from 0 (worst imaginable health) to 100 (best imaginable health).
Pre- and post-operative pain assessment in Urinary Tract Procedure Cohort | From baseline to 6-weeks post procedure
  Pre- and post-operative pain as measured by validated pain questionnaire (Brief Pain Inventory).
Change in uroflowmetry in BPH cohort | Baseline to 12-months after the procedure
  Improvement in uroflowmetry from baseline as measured by change (increase) in maximum urinary flow rate (Qmax) within 12 months of index procedure
Quality of Life for BPH cohort measured by Male Sexual Health Questionnaire (MSHQ) | Baseline to 12-months after the procedure
  Quality of Life for BPH cohort measured via a validated questionnaire, Male Sexual Health Questionnaire (MSHQ). Change in MHSQ score will be assessed. MHSQ score ranges from 0 to 125 with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gita Ghadimi, OD, Study Director — Boston Scientific Corporation
Locations (4):
- United States (4):
  - University of Miami Hospital, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No
Patient data is planned to be summarized in aggregate. Data listings of serious adverse events and any device deficiencies will be reported via anonymized code in clinical study reports as required per local regulations.